CLINICAL TRIAL: NCT00492973
Title: Peri-articular Injections Containing a Corticosteroid During Total Knee Arthroplasty
Brief Title: Do Corticosteroid Injections During Total Knee Replacement Improve Early Clinical Results?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Lexington Clinic (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LCO.2006.2
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis; Post-traumatic; Arthrosis
Keywords: arthroplasty; replacement; knee
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone Acetate; Bupivacaine; Morphine; Epinephrine; Clonidine; Cefuroxime; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients in the active comparator group will receive intraoperative injections containing bupivacaine HCl, morphine, epinephrine, clonidine, cefuroxime, and normal saline, as per the surgeon's standard of care.
  Interventions: Drug: active comparator
- Corticosteroid (Experimental): Patients in the Corticosteroid group will have the same medications as the Control Group with the addition of a corticosteroid (methylprednisolone acetate)
  Interventions: Drug: methylprednisolone acetate

INTERVENTIONS:
Drug: methylprednisolone acetate — Same medications and doses as the active comparator, but with the addition of 40 mg of methylprednisolone acetate
  Arms: Corticosteroid
Drug: active comparator — bupivacaine HCl 80 mg, morphine 4 mg, epinephrine 300 micrograms, clonidine 100 micrograms, cefuroxime 750 mg, and normal saline
  Other Names: bupivacaine HCl; morphine; epinephrine; clonidine; cefuroxime; normal saline
  Arms: Control

SUMMARY:
Prior to surgery, a pharmacist will randomly assign participating patients to one of two groups. One group will get an injection in the knee during surgery that contains medications to limit pain and an antibiotic. A second group will get an injection in the knee during surgery that contains the same pain medications and antibiotic along with a corticosteroid to control inflammation. Corticosteroids are anti-inflammatory medications, not to be confused with muscle-building anabolic steroids you may have heard about in the news. Each patient will have an equal chance of being in either of the two groups. This study will test the safety and efficacy of methylprednisolone acetate in the treatment of pain and inflammation following total knee replacement.

DETAILED DESCRIPTION:
Information collected during your office visits:

The patient will be asked for a brief medical history so that we may determine if the patient can participate in the study. A member of our research team will ask the patient a series of questions about his/her knee. The patient will be asked to answer this series of questions a total of 4 times over the course of 1 year. Also, we will record how well the patient can bend and straighten your knee at these 4 office visits. We will have the patient rate the pain in his/her knee and ask the patient if he/she is satisfied with the surgery. If the patients have any complications, those will also be recorded. The patient will also have X-rays taken of the knee at the postoperative follow-up visits. This is the normal routine following total knee replacement. The X-rays will be read by the surgeon to help determine the success of the surgery.

Injection during total knee replacement surgery:

All patients will receive an injection containing bupivicaine HCl, morphine, epinephrine, clonidine, cefuroxime, and normal saline that will be placed directly into the knee during surgery. In addition, approximately half of the patients in the study will also receive methylprednisolone acetate as part of the injection.

Information being collected during your hospital stay:

During the hospital stay, information will be gathered for this study. A physical therapist will measure how well the patient can bend and straighten the knee. The amount of pain medication that was taken at the hospital will be recorded, and the number of days spent in the hospital will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 95
* Has elected to undergo total knee replacement

Exclusion Criteria:

* Allergy to any of the medications used in the protocol
* History of kidney disease
* Rheumatoid arthritis
* Any systemic conditions associated with chronic pain
* History of deep knee sepsis in the affected extremity
* Unable to understand the questions used to obtain the Knee Society Score
* Minors and prisoners will be excluded from the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Christensen, MD, Principal Investigator — New Lexington Clinic
Locations (1):
- Lexington Clinic Sports Medicine Center, Lexington, Kentucky, United States

REFERENCES:
- [Background] Lombardi AV Jr, Berend KR, Mallory TH, Dodds KL, Adams JB. Soft tissue and intra-articular injection of bupivacaine, epinephrine, and morphine has a beneficial effect after total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):125-30. doi: 10.1097/01.blo.0000147701.24029.cc. PMID 15534532
- [Background] Parvataneni HK, Ranawat AS, Ranawat CS. The use of local periarticular injections in the management of postoperative pain after total hip and knee replacement: a multimodal approach. Instr Course Lect. 2007;56:125-31. PMID 17472300
- [Derived] Christensen CP, Jacobs CA, Jennings HR. Effect of periarticular corticosteroid injections during total knee arthroplasty. A double-blind randomized trial. J Bone Joint Surg Am. 2009 Nov;91(11):2550-5. doi: 10.2106/JBJS.H.01501. PMID 19884426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 5/1/2006 and 5/1/2008, a total of 101 patients were recruited to participate in the study during a regularly-scheduled office visit at an orthopedic clinic.
Pre-assignment Details: Of the 101 patients that were consented, 11 patients opted to cancel surgery, 11 patients asked to be removed from the study prior to surgery, and 3 patients were excluded as they were found to have existing allergies to study medications. The remaining sample of 76 patients were randomly assigned to one of the two study groups.
Groups:
- Control Group: Patients will receive intraoperative injections containing bupivacaine HCl, morphine, epinephrine, clonidine, cefuroxime, and normal saline, as per the surgeon's standard of care.
  active comparator : bupivacaine HCl 80 mg, morphine 4 mg, epinephrine 300 micrograms, clonidine 100 micrograms, cefuroxime 750 mg, and normal saline
- Corticosteroid: Corticosteroid (methylprednisolone acetate)
  methylprednisolone acetate : Same medications and doses as the active comparator, but with the addition of 40 mg of methylprednisolone acetate
Period: Overall Study
Arm/Group | Control Group | Corticosteroid
Started | 37 | 39
Completed | 37 | 38 (One patient died of complications related to deep joint sepsis in the early postoperative period.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Corticosteroid | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 19 | 21 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (11.0) | 65.8 (11.1) | 65.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 7 | 16 | 23
Region of Enrollment [Number; unit: participants]
  United States | 37 | 39 | 76

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Time Frame: days after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Corticosteroid
Number analyzed (Participants) | 37 | 38
days | 3.5 (1.9) | 2.6 (0.7)

2. Primary Outcome: Knee Range of Motion
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Corticosteroid
Number analyzed (Participants) | 37 | 38
degrees | 112.5 (10.3) | 112.4 (12.1)

3. Primary Outcome: Knee Society Scores
Description: The Knee Society Score is on a scale of 0 to 100, with 0 being the worst possible score, and 100 being the best possible score. The Knee Society Score takes into account subjective patient reports of pain and functional ability as well as clinical measures of passive knee range of motion.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Corticosteroid
Number analyzed (Participants) | 37 | 38
units on a scale | 87.1 (11.2) | 83.3 (14.7)

4. Primary Outcome: Amount of Pain Medication Taken Per Day
Time Frame: Average of 3 days after surgery
Measure: Mean (Standard Deviation); unit: mg/day morphine equivalant
Arm/Group | Control Group | Corticosteroid
Number analyzed (Participants) | 37 | 39
mg/day morphine equivalant | 47.8 (35.1) | 46.0 (22.4)

5. Primary Outcome: Patient Satisfaction
Time Frame: 6 weeks, 3 months, and 1 year postoperative
Reporting Status: Not Posted

6. Primary Outcome: Complications, Such as Infections, Hospital Readmissions, Manipulations Under Anesthesia, Etc.
Time Frame: any point during the first postoperative year
Measure: Number; unit: Number of participants with complication
Arm/Group | Control Group | Corticosteroid
Number analyzed (Participants) | 37 | 39
Number of participants with complication | 0 | 3

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: One patient died 25 days after the surgery as a result of complications associated with deep knee joint sepsis. Two other patients underwent manipulation under anesthesia at a mean of 9 weeks after TKA.
Arm/Group | Control Group | Corticosteroid
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/39
Other Adverse Events (participants affected / at risk) | 0/37 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=37) | Corticosteroid (N=39)
Death (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=37) | Corticosteroid (N=39)
Manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
One patient died 25 days after the surgery as a result of complications associated with deep knee joint sepsis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes